CLINICAL TRIAL: NCT00039481
Title: A Phase I Trial Of G3139 (BCL-2 Antisense, NSC# 683428, IND# 58842) Combined With Cytotoxic Chemotherapy In Relapsed Childhood Solid Tumors
Brief Title: Oblimersen Plus Combination Chemotherapy and Dexrazoxane in Treating Children and Adolescents With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01872; ADVL0211; U01CA097452 (NIH); CDR0000069387 (Registry Identifier: PDQ (Physician Data Query)); NCT00061191 (obsolete NCT alias)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac Toxicity; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Cardiotoxicity | interventions — oblimersen; Dexrazoxane; Razoxane; Doxorubicin; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (Oblimersen sodium, cytotoxic chemotherapy) (Experimental): See detailed description.
  Interventions: Biological: oblimersen sodium; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: filgrastim; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: dexrazoxane hydrochloride — Given IV
  Other Names: Cardioxane; Savene; Totect; Zinecard
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of oblimersen plus combination chemotherapy and dexrazoxane in treating children and adolescents who have relapsed or refractory solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of doxorubicin and cyclophosphamide by making the tumor cells more sensitive to the drug. Chemoprotective drugs such as dexrazoxane may protect normal cells from the side effects of chemotherapy

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the dose-limiting toxic effects and recommended phase II dose of oblimersen when combined with cyclophosphamide, doxorubicin, and dexrazoxane in pediatric patients with relapsed or refractory solid tumors.

II. Determine the pharmacokinetic behavior of this regimen in these patients. III. Determine, preliminarily, the antitumor activity of oblimersen in these patients.

IV. Assess the biologic activity of oblimersen in mononuclear cells and tumor tissues, in terms of bcl-2 and related protein expression, in these patients.

OUTLINE: This is a 2-part, multicenter, dose-escalation study.

Part A: Patients receive oblimersen IV continuously on days 1-7. Patients also receive dexrazoxane IV followed by doxorubicin IV over 15 minutes followed by cyclophosphamide IV over 1 hour on days 5 and 6. Filgrastim (G-CSF) is administered subcutaneously once daily beginning on day 8 and continuing until blood counts recover. Treatment repeats every 21 days for up to 18 courses (1 year) in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease whose shortening fraction falls below 28% by echocardiogram or whose total life-time cumulative anthracycline dose exceeds 750 mg/m^2 may receive additional courses of oblimersen and cyclophosphamide without doxorubicin and dexrazoxane.

Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Part B: Patients receive oblimersen at the MTD determined in part A and escalating doses of dexrazoxane, doxorubicin, and cyclophosphamide on the same treatment schedule as in part A.

Cohorts of 3-6 patients receive escalating doses of dexrazoxane, doxorubicin, and cyclophosphamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 12-15 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor at original diagnosis that has failed standard therapy or for which no standard therapy exists

  * Patients must have a disease for which there is no known curative potential
* Patients must meet the following criteria for bone marrow function:

  * Status post stem cell transplantation (SCT)
  * Absolute neutrophil count at least 1,500/mm^3
  * Platelet count at least 100,000/mm^3 (transfusion independent)
  * Hemoglobin at least 8.0 g/dL (RBC transfusions allowed)
* No lymphomas
* No CNS tumors or known metastatic disease to the brain or spinal cord
* Performance status - Karnofsky 50-100% (age 11 to 21)
* Performance status - Lansky 50-100% (age 1 to 10)
* At least 8 weeks
* See Disease Characteristics
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 3 times ULN
* No significant hepatic dysfunction
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Creatinine, based on age, as follows:

  * Age 1 to 5: no greater than 0.8 mg/dL
  * Age 6 to 10: no greater than 1.0 mg/dL
  * Age 11 to 15: no greater than 1.2 mg/dL
  * Age 16 to 21: no greater than 1.5 mg/dL
* No significant renal dysfunction
* Shortening fraction at least 28% by echocardiogram
* Ejection fraction at least 45% by MUGA
* No significant pulmonary dysfunction
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious uncontrolled infections
* No other end-organ dysfunction that would preclude study entry
* No other clinically significant systemic illness
* See Disease Characteristics
* Recovered from prior immunotherapy
* At least 1 week since prior growth factors or other biologic agents
* At least 6 months since prior autologous SCT
* At least 6 months since prior allogeneic bone marrow transplantation and recovered with no evidence of graft-versus-host disease
* No concurrent immunomodulating agents
* No concurrent prophylactic growth factors during the first course of the study
* No concurrent immunotherapy or other biologic therapy
* Recovered from prior chemotherapy
* At least 2 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* No prior life-time cumulative doxorubicin dose of more than 450 mg/m^2 or equivalent
* No other concurrent chemotherapy
* Concurrent chronic steroids allowed
* Recovered from prior radiotherapy
* More than 2 weeks since prior localized palliative radiotherapy (small port)
* More than 6 months since prior substantial radiotherapy to bone marrow (craniospinal radiotherapy, total body irradiation, or hemi-pelvic radiotherapy)
* No concurrent radiotherapy
* Concurrent chronic medications (e.g., narcotics or antiepileptics) allowed
* No other concurrent investigational agents
* No other concurrent cancer therapy

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2002-11; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxic effects and recommended phase II dose, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to day 21
Change in pharmacokinetic behavior of this regimen | Days 1 (pre-infusion), 5, 6, and 8 (end of infusion)
Antitumor activity | Up to day 21
Biologic activity of oblimersen in mononuclear cells and tumor tissues, in terms of B-cell lymphoma 2 (bcl-2) and related protein expression | Up to day 21

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rheingold, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States